CLINICAL TRIAL: NCT06618872
Title: Incremental Diagnostic Value of Tau-PET With [18F]RO948 vs Amyloid-PET in Patients With
Brief Title: Incremental Diagnostic Value of Tau-PET With [18F]RO948 vs Amyloid-PET in Patients With Cognitive Impairment
Acronym: IDV of tau-PET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Valentina Garibotto, Head of Nuclear Medecine and molecular imaging, University Hospital, Geneva
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-02263
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Dementia; Alzheimer Disease
Keywords: Alzheimer; PET; Amyloid; Tau
MeSH Terms: conditions — Dementia; Alzheimer Disease; Pick Disease of the Brain | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: Participants will have first a Tau-PET (experimental) and then an amyloid PET (standard of care) or the opposite
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amyloid-PET and then Tau-PET (Experimental): The participant will have the Amyloid-PET (standard of care) and then Tau-PET (experimental)
  Interventions: Diagnostic Test: PET/CT with RO958 (experimental)
- Tau-PET and then Amyloid-PET (Experimental): The participant will have the Tau-PET (experimental) and then the Amyloid-PET (standard of care)
  Interventions: Diagnostic Test: PET/CT with RO958 (experimental)

INTERVENTIONS:
Diagnostic Test: PET/CT with RO958 (experimental) — the participant will have 2 PET (one with an experimental radiotracer- Tau PET), one with a standard radiotracer (amyloid-PET)

SUMMARY:
The objective of the study is to investigate the clinical validity of tau-PET with [18F]RO948 vs. amyloid-PET in patients with Mild Cognitive Impairment (MCI) or mild dementia

DETAILED DESCRIPTION:
Dementia is defined as cognitive impairment associated with loss of autonomy and is usually preceded by a prodromal phase - Mild Cognitive Impairment (MCI) - which represents a highly heterogeneous entity comprising different underlying etiologies, of which Alzheimer's disease (AD) is one of the most prevalent. Several AD biomarkers - including MRI, FDG-PET and CSF measures of amyloid and tau pathology - have been validated as diagnostic (allowing an early and differential diagnosis of AD) and prognostic (predicting progression from MCI to dementia due to AD) tools. In contrast and despite the increasing consensus on their clinical utility, usage of PET markers of amyloid and tau pathology is not yet standard clinical practice. Moreover, while the clinical utility of amyloid-PET has been exhaustively investigated, to date no study has prospectively assessed the clinical utility of tau-PET. Assessing the clinical utility of diagnostic tools is fundamental for clinical practice. This will be the first study assessing the clinical utility of [18F]RO948 tau-PET vs. standard of care amyloid-PET, providing unique information to define appropriate diagnostic algorithms

ELIGIBILITY:
Inclusion Criteria:

* Written Inform Consent to participating.
* 50 to 85 years of age
* a diagnosis of Mild Cognitive Impairment (MCI=at least one pathological neuropsychological test but no functional impairment based on the Amsterdam IADL score) or mild dementia (both cognitive and functional impairments)
* availability of MRI within 6 months before screening
* prescription of a diagnostic amyloid PET
* Willing and able to comply with the requirements of the study, as judged by the investigator.

Exclusion Criteria:

* The presence of psychiatric disorders, extensive white matter lesions or other stigmata of vascular dementia.
* Visual and auditory acuity inadequate for neuropsychological testing.
* Enrolment in previous clinical trials for AD potentially affecting amyloid and/or tau brain load
* Enrolment in other trials or studies not compatible with [18F]RO948 Imaging study.
* Ferromagnetic implants and devices (including implants or devices held in place by sutures, granulation or ingrowth of tissue, fixation devices, or by other means) not eligible for MRI scanning.
* Women of childbearing potential must not be pregnant (negative urine β-hCG on the day of imaging) or breast feeding at screening

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Difference between tau-PET with [18F]RO948 and amyloid PET in the change of physician's diagnostic confidence (50-100% visual analogue scale) across time | through study completion , an average of 2 years
  Amyloid and tau PET scans will be classified as positive or negative for the presence of pathology using visual reading by an expert reader (amyloid-PET), as clinically established, and SUVR cut offs previously published for [18F]RO948 tau-PET (Leuzy, Smith et al. 2020) as well as a visual check
Difference between tau-PET with [18F]RO948 and amyloid PET in the changes in etiological diagnoses across time (i.e., from Alzheimer disease (AD) to non-AD, or from non-AD to AD). | through study completion , an average of 2 years
  The changes in etiological diagnosis across rounds will be assessed using the McNemar's test

SECONDARY OUTCOMES:
Accuracy of clinical and biomarker-based diagnoses | through study completion , an average of 2 years
  the accuracy of clinical (routine workup only) and biomarker-based diagnoses (based on tau-PET with [18F]RO948 or amyloid-PET or both) using the 2-year follow-up biomarker based diagnosis as gold standard
Amyloid-PET and tau-PET predictivity of cognitive decline and dementia onset | through study completion , an average of 2 years
  The amyloid-PET and tau-PET predictivity of cognitive decline and dementia onset will be assessed using linear mixed models with cognition as dependent variable; results of amyloid-PET or tau-PET, time and their interaction as independent variables; and age, gender and education as covariates
Absence of adverse events | through study completion , an average of 2 years
  Absence of adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Geneva University Hospital, Geneva, Canton of Geneva
  - Centre Medical Universitaire Vaudois, Lausanne, Canton of Vaud

IPD SHARING:
Plan to Share IPD: Undecided